CLINICAL TRIAL: NCT04419818
Title: A Neuropsychological Test Battery for the Assessment of Time Deficits in Brain-damaged Patients: a Correlation Study
Brief Title: A Neuropsychological Test Battery for the Assessment of Time Deficits
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ICS Maugeri CE 2194-Ob2B
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Brain Damage; Health Behavior
Keywords: Time perception; Mental Time Travel; Virtual Reality
MeSH Terms: conditions — Brain Injuries; Health Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Left brain damaged patients: A group of 20 left brain damaged (LBD) patients will perform:
  * a computerized test battery to measure time abilities (Mental Time Travel, Time Estimation and Time Reproduction);
  * a neuropsychological screening (Mini Mental State Examination and Token Test) to assess inclusion/exclusion criteria;
  * questionnaires to evaluate the time needed to execute actions and the ability to locate daily activities in time.
  Interventions: Behavioral: Virtual Reality
- Right brain damaged patients: A group of 20 right brain damaged (RBD) patients will perform:
  * a computerized test battery to measure time abilities (Mental Time Travel, Time Estimation and Time Reproduction);
  * a neuropsychological screening (Mini Mental State Examination and Token Test) to assess inclusion/exclusion criteria;
  * questionnaires to evaluate the time needed to execute actions and the ability to locate daily activities in time.
  Interventions: Behavioral: Virtual Reality
- Healthy controls: A group of 40 (20 young and 20 elderly) healthy controls (HC) will perform:
  * a computerized test battery to measure time abilities (Mental Time Travel, Time Estimation and Time Reproduction);
  * a neuropsychological screening (Mini Mental State Examination) to assess inclusion/exclusion criteria;
  * questionnaires to evaluate the time needed to execute actions and the ability to locate daily activities in time.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — Virtual Reality task consists of a 3D computer-generated virtual environment that will be displayed on a desktop VR computer monitor. A joystick will provide the graphical interface for patients by allowing user-friendly exploration of virtual scenarios. Participants will be presented 16 actions, with dynamic simulations of real life situations. They will verbally estimate and reproduce the duration of each previously presented action.

SUMMARY:
Time processing involves different abilities - i.e. estimating the duration of an event and moving in past and future time - and it is a fundamental ability in everyday life. For these reasons the assessment and the rehabilitation of time deficits in brain damaged patients is extremely important.

The ability to estimate and reproduce time processing is usually evaluated using computerized tasks and it is influenced by aging: young participants overestimate and elderly participants underestimate time durations.

Virtual Reality is an ecological approach that has recently been used for the assessment of cognitive deficits. Here we use Virtual Reality to study the ability to estimate time duration of an action execution and perception in a simulated everyday activity.

DETAILED DESCRIPTION:
Time processing involves different abilities - i.e. estimating the duration of an event and moving in past and future time - and it is a fundamental ability in everyday life. However, in neuropsychology, time processing is routinely neglected in the assessment of cognitive deficits in brain-damaged patients. The discrepancy between the importance of time processing and the lack of instruments for the diagnosis of time deficits in brain damaged patients can be mainly due to the fact that time difficulties fail to emerge in a hospital context where daily activities are routinely scheduled by careers. Thus, time deficits become critical only when patients return home and, for younger patients, when they go back to working activities. For these reasons the assessment and the rehabilitation of time deficits in brain damaged patients is extremely important.

Interestingly, recent evidence has begun to demonstrate that our perceptions and sensations are influenced by motor movements and actions. Further, there is also evidence suggesting that movement not only biases perceived time, but can enhance it, suggesting the motor system directly influences temporal perception.

The ability to estimate and reproduce time in actions is usually evaluated using computerized tasks and it is influenced by aging: young participants overestimate and elderly participants underestimate time durations.

Virtual Reality is an ecological approach that has recently been used for the assessment of cognitive deficits. Here we use Virtual Reality to study the ability to estimate time duration of an action execution and perception in a simulated everyday activity.

The primary aim of the project is to measure the impact of time deficits and its effects on everyday life: a neuropsychological battery assessing time processing (Time Estimation, Time Reproduction, Mental Time Travel) is tested using both computerized and virtual reality tasks.

Moreover, the project aims also to investigate i) the correlation between Time Reproduction in a computerized task and the ability to reproduce the duration of an executed action in Virtual Reality; ii) the correlation between Time Estimation in a computerized task and the ability to estimate the duration of an executed action in Virtual Reality.

ELIGIBILITY:
Inclusion Criteria:

* patients with focal right and left brain-damage

Exclusion Criteria:

* generalized cognitive impairment (score lower than 24 at the Mini Mental State Examination)
* psychiatric disorders
* additional neurological disorders
* abusive use of alcohol or illicit drugs

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from primary care clinic and they will be compared with matched healthy controls. Healthy controls will be selected from a community sample who volunteer to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Assessment of Mental Time Travel Ability on the Mental Time Travel (MTT) Task | baseline
  In the MTT task participants are listened to auditory stimuli consisting of brief descriptions of personal and non-personal events. They are required to project themselves in the past (10 years ago), present or future (10 years from now) and to verbally determine whether each event has already happened (relative past event) or is yet to happen (relative future event) with respect to the specific self-location in time (past, present and future).
  Error rates and reaction times will be recorded and analyzed.
Assessment of Time Estimation Ability on the Time Estimation Task - long intervals | baseline
  The Time Estimation task consists of a red square that is displayed for different durations (3500, 5500, 7500, 9500, 11500 ms) on the computer screen. Participants are instructed to verbally judge whether the duration of each stimulus is "short" or "long" with respect to previously acquired pair of reference durations (3500 and 11500 ms).
  A psychophysical response function will be created for each participant by calculating the proportion of "long" responses: the Point of Subjective Equality (PSE) is the duration at which a participant is equally likely to classify the stimuli as short or long. Lower PSE reflects a relative shift towards overestimation of temporal midpoint. Conversely, higher PSE reflects a relative shift towards underestimation of temporal midpoint.
Assessment of Time Estimation Ability on the Time Estimation Task - short intervals | baseline
  The Time Estimation task consists of a red square that is displayed for different durations (1400, 1700, 2000, 2300, 2600 ms) on the computer screen. Participants are instructed to verbally judge whether the duration of each stimulus is "short" or "long" with respect to previously acquired pair of reference durations (1400 and 2600 ms).
  A psychophysical response function will be created for each participant by calculating the proportion of "long" responses: the Point of Subjective Equality (PSE) is the duration at which a participant is equally likely to classify the stimuli as short or long. Lower PSE reflects a relative shift towards overestimation of temporal midpoint. Conversely, higher PSE reflects a relative shift towards underestimation of temporal midpoint.
Assessment of Time Reproduction Ability on the Time Reproduction Task - long intervals | baseline
  In the Time Reproduction task a blue square is presented for a variable time interval (3500, 5500, 7500, 9500, 11500 ms) on the computer screen. Next, a red square appears on the screen and participants are instructed to reproduce the entire duration of the preceding blue square by pressing the space bar on the keyboard.
  The reproduced time intervals will be compared to the real ones: the difference will be positive when reproduced time will be longer (underestimation of time duration) and negative when reproduced time will be shorter (overestimation of time duration) than the real one.
Assessment of Time Reproduction Ability on the Time Reproduction Task - short intervals | baseline
  In the Time Reproduction task a blue square is presented for a variable time interval (1400, 1700, 2000, 2300, 2600 ms) on the computer screen. Next, a red square appears on the screen and participants are instructed to reproduce the entire duration of the preceding blue square by pressing the space bar on the keyboard.
  The reproduced time intervals will be compared to the real ones: the difference will be positive when reproduced time will be longer (underestimation of time duration) and negative when reproduced time will be shorter (overestimation of time duration) than the real one.

SECONDARY OUTCOMES:
Assessment of Verbal Estimation Ability on the Time and Weight Estimation Test (STEP) | baseline
  The STEP assesses aspects of executive functioning related to cognitive estimation ability. The questionnaire is composed of two distinct ten-item sections, focusing on time (e.g., How long does it take to have a shower?) and weight (e.g., How heavy is a pair of jeans?) estimations. Each item scores from 0 (bizarre estimation) to 3 (best estimation), for a total maximum score for each section of 30, with a cut-off value for normality above 20 for each section.
Assessment of Verbal Estimation Ability on the Cognitive Estimation Task (CET) | baseline
  The test comprised 21 questions requiring participants to give oral, numerical responses. Two different scoring procedures will be considered: absolute error score and bizarreness. The total score for all 21 items ranges from a best of zero to a worst of 42. The greater the error score, the poorer the performance on the CET (cut-off = 18). The total bizarreness score ranges from 0 and 21 (cu-off = 4). The higher the bizarreness score, the greater the impairment in cognitive estimation.
Assessment of Functional Abilities on the Questionnaire of Temporal Ability | baseline
  The Questionnaire of temporal ability is a new instrument to measure the ability to locate 10 daily activities in time.
Assessment of General Cognitive Functioning on the Mini Mental State Examination (MMSE) | baseline
  The MMSE is a 30-point questionnaire that examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. The score ranges from 0 to 30 (cut-off = 24).
Assessment of Verbal Comprehension on the Token Test | baseline
  The Token test is a test of auditory language processing in which participants are asked to manipulate tokens of different shapes, sizes, and colors in response to increasingly complex instructions. One point is credited for a correct performance on the first presentation and 0.5 point if the performance is correct only on the second presentation. The score ranges from 0 to 36 (cut-off = 26,50).
Correlation between Time Estimation, Time Reproduction and Virtual Reality | baseline
  Time Estimation, Time Reproduction and VR tasks will be correlated to investigate the relationship between computerized tasks and virtual reality tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Frassinetti, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri IRCCS
Locations (1):
- ICS Maugeri IRCCS, U.O. di Rieducazione e Recupero funzionale di Castel Goffredo, Castel Goffredo, Mantova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anelli F, Avanzi S, Arzy S, Mancuso M, Frassinetti F. Effects of spatial attention on mental time travel in patients with neglect. Cortex. 2018 Apr;101:192-205. doi: 10.1016/j.cortex.2018.01.012. Epub 2018 Feb 2. PMID 29482017
- [Background] Anelli F, Avanzi S, Damora A, Mancuso M, Frassinetti F. Mental time travel and functional daily life activities in neglect patients: Recovery effects of rehabilitation by prism adaptation. Cortex. 2019 Apr;113:141-155. doi: 10.1016/j.cortex.2018.12.003. Epub 2018 Dec 14. PMID 30660953
- [Background] De Renzi E, Faglioni P. Normative data and screening power of a shortened version of the Token Test. Cortex. 1978 Mar;14(1):41-9. doi: 10.1016/s0010-9452(78)80006-9. PMID 16295108
- [Background] Della Sala S, MacPherson SE, Phillips LH, Sacco L, Spinnler H. How many camels are there in Italy? Cognitive estimates standardised on the Italian population. Neurol Sci. 2003 Apr;24(1):10-5. doi: 10.1007/s100720300015. PMID 12754651
- [Background] Demeurisse G, Demol O, Robaye E. Motor evaluation in vascular hemiplegia. Eur Neurol. 1980;19(6):382-9. doi: 10.1159/000115178. PMID 7439211
- [Background] Espinosa-Fernandez L, Miro E, Cano M, Buela-Casal G. Age-related changes and gender differences in time estimation. Acta Psychol (Amst). 2003 Mar;112(3):221-32. doi: 10.1016/s0001-6918(02)00093-8. PMID 12595147
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Frassinetti F, Magnani B, Oliveri M. Prismatic lenses shift time perception. Psychol Sci. 2009 Aug;20(8):949-54. doi: 10.1111/j.1467-9280.2009.02390.x. Epub 2009 Jun 22. PMID 19549081
- [Background] Patane I, Farne A, Frassinetti F. Prismatic Adaptation Induces Plastic Changes onto Spatial and Temporal Domains in Near and Far Space. Neural Plast. 2016;2016:3495075. doi: 10.1155/2016/3495075. Epub 2016 Feb 14. PMID 26981286
- [Background] Wiener M, Zhou W, Bader F, Joiner WM. Movement Improves the Quality of Temporal Perception and Decision-Making. eNeuro. 2019 Aug 20;6(4):ENEURO.0042-19.2019. doi: 10.1523/ENEURO.0042-19.2019. Print 2019 Jul/Aug. PMID 31395616
- [Result] Cantarella G, Vianello G, Vezzadini G, Frassinetti F, Ciaramelli E, Candini M. Time bisection and reproduction: Evidence for a slowdown of the internal clock in right brain damaged patients. Cortex. 2023 Oct;167:303-317. doi: 10.1016/j.cortex.2023.05.024. Epub 2023 Jul 25. PMID 37595392